CLINICAL TRIAL: NCT06978322
Title: Comparative Study Between Immediate Surgery Versus Neoadjuvant Chemotherapy for Management of Resectable Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer of General Surgery, Faculty of Medicine, Minia University, Minia, Egypt., Minia University
Other Study IDs: 1437/02/2025
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Neoadjuvant Chemotherapy; Management; Resectable Pancreatic Cancer
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate surgery group: Patients will undergo upfront surgery, then adjuvant chemotherapy.
  Interventions: Procedure: Immediate surgery
- Neoadjuvant chemotherapy group: Patients will undergo neoadjuvant chemotherapy, then surgery.
  Interventions: Procedure: Neoadjuvant chemotherapy

INTERVENTIONS:
Procedure: Immediate surgery — Patients will undergo upfront surgery, then adjuvant chemotherapy.
  Groups: Immediate surgery group
Procedure: Neoadjuvant chemotherapy — Patients will undergo neoadjuvant chemotherapy, then surgery.
  Groups: Neoadjuvant chemotherapy group

SUMMARY:
This trial aimed to determine whether neoadjuvant chemoradiotherapy improves overall survival compared with upfront surgery, both followed by adjuvant chemotherapy in patients with resectable and borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the solid cancers with the poorest treatment outcomes, and there is an urgent need to improve its treatment outcomes. Among these, resectable pancreatic cancer is known to show relatively good treatment outcomes with surgical resection, but the 5-year survival rate is still about 20%, which is still unsatisfactory.

Neoadjuvant therapy may increase the proportion of patients that actually receive chemotherapy and thereby improve survival. Furthermore, neoadjuvant therapy may increase the microscopically margin-negative (R0) resection rate and may identify patients with rapidly progressive disease who can be spared futile surgery.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography (CT) with pancreatic protocol + vascular mapping
* Histopathologically proven malignant by CT-guided or endoscopic ultrasound (EUS)-guided biopsy Resectable pancreatic cancer means no contact of the tumor with the Superior mesenteric artery, Celiac axis & Common hepatic artery, and contact of the tumor but ≤90° contact with the superior mesenteric vein & portal vein.

Exclusion Criteria:

* Borderline resectable & locally advanced pancreatic cancer
* Tumor at the tail of the pancreas.
* Metastatic pancreatic cancer
* Unfit patients for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective and retrospective study will be conducted on 30 patients with resectable pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 1 year post-procedure
  Overall survival will be measured as the time between date of randomization and date of death from any cause or date of last follow-up if alive.

SECONDARY OUTCOMES:
Achieve of R0 Resection | 1 year post-procedure
  Resection is defined as the number of patients with an R0 resection margin. R0 resection margin rate will be measured according to the Africa Regional Collaborative Platform (RCP) report on standards and datasets for reporting cancers.
Disease free survival | 1 year post-procedure
  Disease-free survival will be measured as the time between date of surgery and date of disease recurrence.
Time to locoregional recurrence | 1 year post-procedure
  Time to locoregional recurrence will be recorded.
Time to distant metastasis | 1 year post-procedure
  Time to distant metastasis will be recorded.
Incidence of postoperative complications | 1 year post-procedure
  Incidence of postoperative complications such as hemorrhage and pancreatic fistula will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.